CLINICAL TRIAL: NCT04604912
Title: Multi-omics Endotyping of Food-allergic Patients For Advanced Biomarker Discovery
Brief Title: Biomarkers in Food Allergy Diagnosis
Acronym: APSIS
Status: Completed | Type: Observational
Sponsor: Luxembourg Institute of Health (Other Government)
Collaborators: Centre Hospitalier du Luxembourg (Other); Odense University Hospital (Other); Technical University of Munich (Other); University of Luxembourg (Other); Integrated Biobank of Luxembourg (Other)
Responsible Party: Sponsor
Other Study IDs: APSIS
Record Dates: First submitted 2020-09-30; First posted 2020-10-27 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Allergy;Food
Keywords: Peanut allergy; Active peptides; Oral food challenge; Immune cell phenotyping; Microbiome
MeSH Terms: conditions — Food Hypersensitivity; Peanut Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Blood-derived samples (sera, plasma, peripheral blood mononuclear cell/PBMC) and stool will be collected
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Peanut-allergic patients' group: The aim is to include 30 patients with peanut allergy. Those patients will undergo diagnostic food challenges (incremental doses) while blood will be samples before, during and after the testing. The patients will receive standard of care during and after the challenge. Allergic symptoms will be treated according to established guidelines.
- Control group: The aim is to include 20 control participants, 10 peanut-tolerant and 10 fish-tolerant individuals. Those participants will undergo diagnostic food challenges (incremental or single doses) while blood will be samples before, during and after the testing. Same safety measures will be applied for food challenges of control individuals, as for the allergic patients.

SUMMARY:
Food allergy is a global burden, affecting patients, society as a whole and the economy. For most common food allergies, patients synthesize specific IgE-antibodies against harmless food proteins. Clinical phenotypes of food-allergic patients are highly diverse. Differences in medical symptoms (organs, severity, delay), threshold and cross-reactivity levels suggest variable underlying endotypes.

The aim of this study is to identify phenotypic biomarkers for advanced stratification of food-allergic patients. Our study will consist of up to 50 participants (30 food-allergic, 20 tolerant), recruited in Luxembourg. Clinical samples will be collected before, during and after the event of a double-blind placebo-controlled food challenge for patients. Multi-omics analyses of blood (sera, peripheral blood mononuclear cell, basophils) and stool will allow a deeper understanding of the underlying immune mechanisms, including allergen metabolism aspects, as well as the functional gut microbiome. Deciphering these basic aspects during the present pilot study is expected to pave the way towards novel personalized medicine approaches for diagnosing and treating of food-allergic individuals.

This study is a cooperation project between the Centre Hospitalier de Luxembourg (CHL), the Luxemburg Institute of Health (LIH), the University of Luxembourg and the Integrated Biobank of Luxemburg (IBBL).

DETAILED DESCRIPTION:
Background. Food allergies are a global burden causing severe clinical reactions including fatal anaphylaxis. Peanuts are counted among the most potent elicitors involved in IgE-mediated food allergies. Peanut allergy is a relevant disease model because of its steadily increasing prevalence and poor prognosis of outgrowth. Clinical phenotypes of peanut-allergic patients are highly variable. Patients might experience variable medical symptoms (organs, severity, delay), threshold and cross-reactivity levels suggest. Reliable in-vitro biomarker allowing to predict clinical reactivity and score the patients into reaction endotypes are missing.

Most important peanut allergens have been studied as to their biomolecular properties biological activities and allergenic potency. The pronounced protein stability of potent peanut allergens is thought to contribute to the molecules' allergenicity. Upon ingestion, food proteins are broken down, entering the human body via epithelial surfaces. The identity and the fate of immunologically active allergen peptides after epithelial absorption remains elusive. Beyond this, complex immune cascades take place during acute allergic episodes. How immune cells, such as lymphocytes, orchestrate in patients with different clinical outcomes (e.g., sensitivity, severity) still remains to be solved. Several studies have shown that the composition and the diversity of the gut microbiota is relevant for shaping the immune response to food proteins. The functional interaction between host and gut microbiome, in the context of symptom development and phenotypic variations, is unexplored until today.

Aims. This project aims to explore putative biomarkers at various levels, at the level of IgE-profiles, at the level of allergen absorption, at the level of scored basophil reactivity, at the level of immune phenotypes and at the level of gut microbiome-host interactions, by applying multiple omics technologies.

Partners. The Luxembourg Institute of Health (LIH), Department of Infection and Immunity (DII; head Prof. M. Ollert) has the scientific project lead (Principal Investigator Dr. A. Kuehn). Main clinical partners are Dr. F. Codreanu-Morel from the National Unit of Immunology-Allergology, Centre Hospitalier (CHL), Luxembourg, as well as Prof. C. Bindslev-Jensen from Odense Research Centre for Anaphylaxis (ORCA), Denmark. Partner for the execution of the clinical part will be the Clinical and Epidemiological Investigation Center (CIEC, LIH) headed by Dr. M. Gantenbein. The Integrated Biobank of Luxembourg (IBBL) will prepare and store clinical samples until use. Clinical samples (blood, sera, plasma) will be analyzed at DII, LIH. Stool samples will be investigated with the help of Prof. P. Wilmes from the Systems Ecology research group, Luxembourg Centre for Systems Biomedicine (LCSB).

Project implementation. Food challenges (OFC) to peanut will be proceeded according to official guidelines (European Academy of Allergy and Clinical Immunology, EAACI). Healthy controls (N=10) will be split, half will receive a single food dose of up to 100 g of roasted peanuts (open OFC) and the other half will be tested with up to 5 incremental doses (double-blind placebo-controlled OFC) using the same doses as for allergic patients. For single-dose OFC, blood samples from controls will be taken before the OFC and at 30 minutes, at 60 minutes and at 120 minutes. Controls receiving 5 incremental allergen doses will be subjected to blood sampling before the beginning of the OFC and 1 h after the end of the challenge. As a further control arm in the study, allergenic food from animal origin will be used in OFC. Further healthy controls (N=10) will receive either a single food dose of up to 200 g of cooked fish (open OFC) and the other half will be tested with up to 5 incremental doses (double-blind placebo-controlled OFC). Doses in a range of 10 mg to 100 g of fish will be selected for the blinded OFC with controls.

Allergic participants (N=30) will ingest incremental doses of peanuts. The OFC doses will be in the range of 5 mg, 15 mg, 60 mg, 120 mg, 200 mg, 390 mg, 790 mg, 1,580 mg, 3,160 mg and 5,530 mg of roasted peanut. Maximum five doses will be selected from the above mentioned ranges of peanut doses. Upon observation of allergic symptoms, the OFC will be stopped. If no allergic symptoms occurred during a food challenge with five incremental doses, the patient will be asked to participate in a second oral provocation (min. 14 days later) in order to undergo a test with higher allergen doses. Blood samples from allergic study participants will be drawn prior, during and after OFC (0, 60, 150, 180 minutes).

Stool samples from peanut-allergic participants (n=30) and healthy controls (n=20) will be collected earliest 2 months after the food challenge. Prior sampling, participants should not have used antibiotics within the last month, or have recent/ongoing gastrointestinal symptoms (= diarrhea; Bristol scale 5-7) at the time of stool collection. Participants will receive a collection kit at home, containing special sampling tubes, gloves and instructions. In addition, patients are asked to record their food intake for the last 24 hours before sampling.

Collected clinical samples will be pseudonymized at the clinical centers. A synonym list, as part of the investigator file, containing the information on the participants' identity and the corresponding pseudonym, will be available at the clinical center only (medical investigators) and at CIEC. Personal data is protected under the regulation (EU) 2016/679 of 27 April 2016 on the protection of individuals with regard to the processing of personal data (GDPR) and the law of 1 August 2018 on the organization of the National Data Protection Commission and the General Data Protection Act.

ELIGIBILITY:
For the allergic cohort :

Inclusion criteria:

* 2-70 years
* male or female
* Allergic to peanut (assessed by anamnesis, skinreactivity testing, sera testing for specific IgE)
* Sign an Informed Consent
* Diagnostic food challenge scheduled

Exclusion criteria:

* Significant co-morbidity
* Medical treatment by nonsteroidal anti-inflammatory drugs oraspirin, chronic treatment with beta-blockers,angiotensin-converting enzyme inhibitors, use ofantihistamines within 5 days of oral food challenge and oral corticosteroids within 14 days prior to the challenge
* Medical unfit for challenge (e.g : fever,unwell with intercurrent illness)
* Pregant women
* Unbalanced asthma
* Severe food-induced anaphylaxis

For the control cohort :

Inclusion criteria:

* Adults
* male or female
* Sign an Informed Consent
* Tolerance to peanuts and fish (IgE-titer < 0.10 kUA/L)

Exclusion criteria

* Pregnancy
* Medical unfit for challenge (e.g : fever, unwell with intercurrent illness),
* Unbalanced asthma
* Treatment by nonsteroidal anti-inflammatory drugs or aspirin
* Chronic treatment with beta-blockers, angiotensin-converting enzyme inhibitors
* Use of antihistamines within 5 days of oral food challenge
* Oral corticosteroids within 14 days prior to the challenge
* Risk of severe food-induced anaphylaxis in highly sensitized peanut-allergic patients

Ages: 2 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Peanut-allergic individuals (N=30) and tolerant controls (N=20). Among the allergic patients, up to 10 allergic individuals of age 2-5 will be included.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in peripheral allergen peptides (serum samples) across food allergen uptake | Samples analyzed through study completion, an average of 3 months
  Abundance of allergen peptides as detected through mass spectrometry. Main comparison will be on two study arms, food-allergic patients versus healthy controls
Change in in-vitro basophil reactivity profiles (cells sampled before food challenge) using defined food allergen peptides across different peptides mixes and peptide concentrations | Samples analyzed through study completion, an average of 3 months
  Reactivity of effector cells by dose-dependent activation (%-CD63+ CCR3+basophils) and flow cytometry measurement. Main comparison will be within the group of food-allergic patients, aligning patients with high/low reactivity and high/low sensitivity of basophils.
Change of immune cell phenotypes across food allergen uptake | Samples analyzed through study completion, an average of 3 months
  Abundance and function of immune cells as detected through single-cell mass cytometry. Main comparison will be on two study arms, food-allergic patients versus healthy controls.
Change in Cytokine release | Samples analyzed through study completion, an average of 3 months
  Cytokine quantification through multiplex immunoassays. Main comparison will be on two study arms, food-allergic patients versus healthy controls.
Baseline characteristics of the functional gut microbiome in food-allergic patients | Samples analyzed through study completion, an average of 2 months
  DNA, RNA, protein and metabolite profiling using a multi-omics approach through 16S RNA sequencing, unbiased high resolution method of metagenomics shotgun sequencing and transcriptomic analysis (Illumina MiSeq & NextSeq) as well as metabolomic analysis (gas chromatography-mass spectrometry/liquid chromatography-mass spectrometry). In addition, microbial component analysis by antibody-specific immunoassays and flow cytometry. Main comparison will be on two study arms, food-allergic patients versus healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Annette Kuehn, PhD, Principal Investigator — Luxembourg Institute of Health
Locations (2):
- Luxembourg (2):
  - Luxembourg Institute of Health, Esch-sur-Alzette
  - Centre Hospitalier Luxembourg, Luxembourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Muraro A, Lemanske RF Jr, Castells M, Torres MJ, Khan D, Simon HU, Bindslev-Jensen C, Burks W, Poulsen LK, Sampson HA, Worm M, Nadeau KC. Precision medicine in allergic disease-food allergy, drug allergy, and anaphylaxis-PRACTALL document of the European Academy of Allergy and Clinical Immunology and the American Academy of Allergy, Asthma and Immunology. Allergy. 2017 Jul;72(7):1006-1021. doi: 10.1111/all.13132. Epub 2017 Apr 12. PMID 28122115
- [Background] Matricardi PM, Kleine-Tebbe J, Hoffmann HJ, Valenta R, Hilger C, Hofmaier S, Aalberse RC, Agache I, Asero R, Ballmer-Weber B, Barber D, Beyer K, Biedermann T, Bilo MB, Blank S, Bohle B, Bosshard PP, Breiteneder H, Brough HA, Caraballo L, Caubet JC, Crameri R, Davies JM, Douladiris N, Ebisawa M, EIgenmann PA, Fernandez-Rivas M, Ferreira F, Gadermaier G, Glatz M, Hamilton RG, Hawranek T, Hellings P, Hoffmann-Sommergruber K, Jakob T, Jappe U, Jutel M, Kamath SD, Knol EF, Korosec P, Kuehn A, Lack G, Lopata AL, Makela M, Morisset M, Niederberger V, Nowak-Wegrzyn AH, Papadopoulos NG, Pastorello EA, Pauli G, Platts-Mills T, Posa D, Poulsen LK, Raulf M, Sastre J, Scala E, Schmid JM, Schmid-Grendelmeier P, van Hage M, van Ree R, Vieths S, Weber R, Wickman M, Muraro A, Ollert M. EAACI Molecular Allergology User's Guide. Pediatr Allergy Immunol. 2016 May;27 Suppl 23:1-250. doi: 10.1111/pai.12563. PMID 27288833
- [Background] Bunyavanich S, Berin MC. Food allergy and the microbiome: Current understandings and future directions. J Allergy Clin Immunol. 2019 Dec;144(6):1468-1477. doi: 10.1016/j.jaci.2019.10.019. PMID 31812181
- [Background] Costa J, Bavaro SL, Benede S, Diaz-Perales A, Bueno-Diaz C, Gelencser E, Klueber J, Larre C, Lozano-Ojalvo D, Lupi R, Mafra I, Mazzucchelli G, Molina E, Monaci L, Martin-Pedraza L, Piras C, Rodrigues PM, Roncada P, Schrama D, Cirkovic-Velickovic T, Verhoeckx K, Villa C, Kuehn A, Hoffmann-Sommergruber K, Holzhauser T. Are Physicochemical Properties Shaping the Allergenic Potency of Plant Allergens? Clin Rev Allergy Immunol. 2022 Feb;62(1):37-63. doi: 10.1007/s12016-020-08810-9. PMID 32876924
- [Background] Jappe U and Kuehn A. Neues zu diagnostisch relevanten Einzelallergenen aus pflanzlichen und tierischen Nahrungsmittelallergenquellen. Allergologie 2016; 39: 425-438. doi: 10.5414/ALX01885.